CLINICAL TRIAL: NCT03786536
Title: Clinical Investigation of the Safety and Initial Performance of the MediSieve Magnetic Haemofiltration System in Healthy Volunteers
Brief Title: Safety and Initial Performance of the MediSieve Magnetic Haemofiltration System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Approval of specific study by UK MHRA not received. Study performed in different circumstances and with different clinical sites / partners.
Sponsor: MediSieve Limited (Industry)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSV_2018/01
Record Dates: First submitted 2018-11-29; First posted 2018-12-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Haemofiltration

STUDY DESIGN:
Intervention Model Description: Healthy volunteer study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All volunteers will receive the same treatment
  Interventions: Device: MediSieve Magnetic Haemofiltration System

INTERVENTIONS:
Device: MediSieve Magnetic Haemofiltration System — The MediSieve Magnetic Haemofiltration System is a medical device intended for use in extracorporeal clinical procedures to remove magnetic targets (e.g. malaria infected red blood cells) from a patient's bloodstream.

SUMMARY:
This is a single centre, prospective, non-randomised healthy volunteer study to be undertaken at University College Hospital London.

The study will be used to demonstrate the safe use of the MediSieve blood filtration system in healthy volunteers prior to undertaking clinical trials on patients with relevant pathologies.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers who meet the following criteria will be considered eligible for the study:

1. Male or female, at least 18 and ≤30 years of age;
2. Able to comprehend and sign the Informed Consent prior to enrolment in the study.

Exclusion Criteria:

Volunteers who meet the following criteria will NOT be eligible for the study:

1. Aged <18 years of age;
2. Aged >30 years of age;
3. Pregnant or lactating females;
4. Individuals < 50kg
5. Individuals with an Hb blood level below 115 g/L
6. Individuals with coagulopathies or under medication that affects normal blood coagulation profile, including COCP in females;
7. Individuals with a previous history of heparin-induced thrombocytopenia;
8. Individuals with known allergy to heparin;
9. Individuals with acute or chronic concomitant conditions; such as diabetes, hypertension, autoimmune disease requiring on going therapy
10. Individuals with history of cancer in the last 5 years;(excluding localised skin cancer or CIS)
11. Individuals with haemoglobinopathy disease;
12. Concurrent participation in another experimental intervention or drug study;
13. Unwilling or unable to provide informed consent.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability, measured by incidence of Treatment-Emergent Adverse Events. | During the study duration of 2 months and within the 6 month time period following treatment with the study device. following treatment
  Treatment-Emergent Adverse Events during the study and the 6 month period after volunteers exit the study. Definitions from ISO14155 will be used to categorise Adverse Events

SECONDARY OUTCOMES:
Performance of device during use. Time required for the user to set up and shut down the haemofiltration pump.. | Through study completion, an average of 6 months...
  Set up and shut down duration. The time, in minutes, to set up and shut down the haemofiltration pump will be recorded for each participant..
Performance of device during use will be assessed by the incidence of flow-rate alarms on the haemofiltration pump during use. | Through study completion, an average of 6 months
  Device performance will be assessed by the incidence of alarms on the haemofiltration pump that are triggered by blood flow through the pump falling below pre-set level..

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Blanco Andujar, PhD, Study Director — MediSieve Limited

IPD SHARING:
Plan to Share IPD: Undecided